CLINICAL TRIAL: NCT01768468
Title: Double Blinded, Randomized, Active Drug Comparative, Multi-center, Phase IV Clinical Study to Compare the Efficacy and Safety of LAYLA in Osteoarthritis Patients
Brief Title: To Compare the Efficacy and Safety of LAYLA in Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PMG Pharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAYLA-P4
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: LAYLA; Non-inferiority; 100mm pain VAS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAYLA (Experimental): Drug : LAYLA tablet/ bid
  Interventions: Drug: LAYLA tablet
- JOINS (Active Comparator): Drug : JOINS tablet/ tid
  Interventions: Drug: JOINS tablet

INTERVENTIONS:
Drug: LAYLA tablet — 1 tablet twice a day
  Other Names: LAYLA 405.4mg
  Arms: LAYLA
Drug: JOINS tablet — 1 tablet at each time, 3 times a day
  Other Names: JOINS 200mg
  Arms: JOINS

SUMMARY:
This is a randomized, double-blind study to compare the efficacy and safety of LAYLA tablet and Joins tablet in the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 and ≤ 80years of age
* Radiographic evidence of grade 2 or 3 osteoarthritis based on the Kellgren & Lawrene radiographic entry criteria
* Stable osteoarthritis during 3 months
* Score of 100mm pain VAS ≤ 80mm at screening
* Score of 100mm pain VAS ≥ 50mm at baseline
* Written consent form voluntarily

Exclusion Criteria:

* Disease of spine or other Lower limb joints that could affect to evaluate the efficacy
* History of surgery or arthroscopy of the study joint within 6 months
* Trauma of study joint within 12 months
* Medication of constantly(more than 1 week) corticosteroid by oral within 3 months
* Medication of intra-articular injection within 3 months
* Diagnosed with psychical disorder, and taking medication
* History of upper gastrointestinal ulceration within 6 months
* History of upper gastrointestinal bleeding within 12 months
* Serum creatinine, ALT, AST, total bilirubin over UNL X 2.0 at screening test
* History of hypersensitivity to LAYLA, JOINS, or NSAIDs
* Participation in another clinical trials within 4 weeks
* Medication of constantly (more than 1 week) narcotic analgesics within 3 months
* Not consent about using effectual contraception method during trial
* Pregnant or lactating woman
* Investigator's judgment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in 100mm Pain VAS | baseline throgh week 8

SECONDARY OUTCOMES:
Change from baseline in 100mm pain VAS | 12 weeks
Change rate from baseline in 100mm Pain VAS | 8 weeks, 12 weeks
Change from baseline in WOMAC | 8 weeks, 12 weeks
Change from baseline in EQ-5D | 8 weeks, 12 weeks
Change in the patient self-assessed & investigator-assessed overall symptom score | 8 weeks, 12 weeks
Consumption of rescue medication | 4 times

CONTACTS AND LOCATIONS:
Overall Officials: Ye Soo Park, Principal Investigator — Hanyang University Guri Hospital; Chul Won Ha, Principal Investigator — Samsung Medical Center; Ye Yeon Won, Principal Investigator — Ajou University School of Medicine; Jae Hyup Lee, Principal Investigator — SMG-SNU Boramae Medical Center; Byung Woo Min, Principal Investigator — Keimyug University Dongsan Medical Center; Seung Beom Han, Principal Investigator — Korea University Anam Hospital
Locations (6):
- South Korea (6):
  - Keimyug University Dongsan Medical Center, Daegu
  - Hanyang University Guri Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Ha CW, Park YB, Min BW, Han SB, Lee JH, Won YY, Park YS. Prospective, randomized, double-blinded, double-dummy and multicenter phase IV clinical study comparing the efficacy and safety of PG201 (Layla) and SKI306X in patients with osteoarthritis. J Ethnopharmacol. 2016 Apr 2;181:1-7. doi: 10.1016/j.jep.2016.01.029. Epub 2016 Jan 25. PMID 26821189